CLINICAL TRIAL: NCT02114034
Title: Cohort Analysis of Clinical and Biological Severe Childhood Asthma
Acronym: COBRAPed
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI12004; N° ID RCB: 2012-A00539-34
Record Dates: First submitted 2013-08-22; First posted 2014-04-15 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Severe Asthma
Keywords: Severe asthma,; child,; outcome,
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * whole blood
  * serum
  * Bronchoalveolar lavage fluid
  * bronchial brushing and washing specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-severe asthma: * Children Controlled without treatment or with low doses of inhaled corticosteroids (<500 mg / day beclometasone equivalent) asthma
  * and Children with normal EFR
  * and Children who did not have more severe exacerbation (assessed taking oral corticosteroids) in the previous year
  * and Children not admitted in the previous year for asthma
- Severe asthma: Asthmatic child who, despite treatment with a combination of inhaled corticosteroids (at least 800 mcg / day equivalent Beclomethasone) bronchodilators and long-acting or properly taken daily leukotriene (inhaler technique and compliance verified) presents one of the 3 criteria following:
  * Persistence of symptoms or chronic use of bronchodilators short duration of action at least three times a week for at least 3 months
  * exacerbations in the previous year:
    * at least one care unit admission or continued resuscitation
    * at least two hospitalizations for acute severe asthma requiring IV therapy
    * at least 2 courses of oral corticosteroids for exacerbations
  * post BD FEV <80% or UARS post BD> 150% predicted

SUMMARY:
The purpose of this prospective study is:

* to identify by cluster analysis the main phenotypes of severe asthma and factors involved in the severity,
* to determine the clinical and functional outcomes,
* to identify the factors associated with severe asthma from childhood to adulthood.

DETAILED DESCRIPTION:
Severe asthma involves about 5 % of asthmatic children and is associated with a high impact on hospitalizations, absenteeism and quality of life.

Although our knowledge has progressed in a substantial way during the last ten years, a number of unresolved questions persist in particular as regard to the contributing factors and outcomes from early childhood to adulthood.

After parental agreement the following elements will be collected at inclusion: clinical environmental data, pulmonary function, allergy test data (skin prick tests and specific IgE), blood and serum samples for biobank (DNA / SERUM). In a restricted number of children a more extensive work up will be performed which may include flexible bronchoscopy, bronchial brushing and bronchoalveolar lavage.

The follow-up will be performed every 6 months within the framework of the usual care including collection of clinical data and pulmonary function tests. The allergic status will be done again at 6-7 years, 12 years and 18 years.

In the group of children having non-severe asthma, the follow-up will be annual with collection of clinical data and pulmonary function tests.

ELIGIBILITY:
Inclusion Criteria:

Children with severe asthma:

* Child aged 3 to 12 years
* Asthmatic child who, despite treatment with a combination of inhaled corticosteroids (at least 800 mcg / day equivalent Beclomethasone) bronchodilators and long-acting or properly taken daily leukotriene or short acting nebulized bronchodilators (inhaler technique and compliance verified) presents one of the criteria following:
* Persistence of symptoms or chronic use of bronchodilators short duration of action at least three times a week for at least 3 months
* exacerbations in the previous year:

  * at least one care unit admission or continued resuscitation
  * at least two hospitalizations for acute severe asthma requiring IV therapy
  * at least 2 courses of oral corticosteroids for exacerbations
* post BD FEV <80% or UARS post BD> 150% predicted
* Signature of consent or the holder (s) of parental authority
* Particular case of patients treated with Xolair® : Patients currently receiving Xolair® but who met the severity criteria of asthma, as described above, before the start of treatment with Xolair® are includable.

Children with non-severe asthma:

Inclusion Criteria

* Child aged 3 to 12 years
* Controlled without treatment or with low doses of inhaled corticosteroids (<500 mg / day beclometasone equivalent) asthma
* Child with normal EFR (Child over 4 years)
* Child who did not have more severe exacerbation (assessed taking oral corticosteroids) in the previous year
* Child not admitted in the previous year for asthma.
* Signature of consent or the holder (s) of parental authority

Exclusion Criteria:

* Child with bronchopulmonary dysplasia
* Child with severe sequelae of viral infections
* Refusal of the child or parents Data collection for research and follow up of patients : tests carried out in the 3 months prior to inclusion are used

Blood sample for DNA extraction and the biobank: for young children, sampling at least 4 to 5 ml on dry tubes for serum and 6 ml at least for DNA. These samples should be stored at room temperature, transported within 48 hours to biological resources (CRB) Necker E,fa,ts Malades.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
The identification of risk factors for severe asthma | 18 years
  A prospective follow-up of a cohort of severe pediatric asthma. To improve the identification of risk factors for severe asthma, a group of children with non-severe asthma will also be included

SECONDARY OUTCOMES:
In the medium and longer term assessment | 4 years
  * Identify the functional and clinical outcome in a longitudinal follow-up to a link with asthma in adults.
  * Identify the factors involved appearing during growth or adulthood (pediatric factors associated with severe asthma profile adult).
A short-term assessment | 4 years
  * Identify the main phenotypes of severe asthma by the cluster analysis
  * Identify the factors involved in severity during childhood
Establish a collection of biological samples (serum bank, DNA Bank, tissue Bank) to search for biomarkers of severity and genetic risk factors for the development of asthma in children. | 18 years

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LEZMI, MD, PhD, Principal Investigator — Assistance Publique-Hôpitaux Paris
Locations (1):
- Service de Pneumologie et allergologie pédiatrique, Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lezmi G, Lejeune S, Pin I, Blanchon S, Bouazza N, Jolaine V, Marguet C, Houdoin V, Berger P, Fayon M, Dubus JC, Reix P, Pellan M, Brouard J, Chiron R, Giovannini-Chami L, Deschildre A, de Blic J; COBRAPed Study Group. Factors Associated with Asthma Severity in Children: Data from the French COBRAPed Cohort. J Allergy Clin Immunol Pract. 2021 May;9(5):1969-1979. doi: 10.1016/j.jaip.2020.12.027. Epub 2020 Dec 24. PMID 33359443